CLINICAL TRIAL: NCT06131528
Title: Effects of Relaxation Breathing Exercises on Cardiovascular Parameters Among Hypertensive Patients
Brief Title: Relaxation Breathing Exercises Effects Among Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Rida Ali
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
Keywords: Relaxation Breathing Exercise; Cardiovascular parameters; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation Breathing Exercises Group (Experimental): This group preformed Relaxation Breathing Exercises that includes Slow Deep Breathing, Pursed lip Breathing, Deep Diaphragmatic Breathing and Alternate Nostril Breathing on alternative pattern for 10 minutes to 30 minutes. These exercises are performed daily with 6 breaths per min. The minimum duration was 3 min for one session.
  Interventions: Other: Relaxation Breathing Exercises Group
- Usual Care Group (Active Comparator): The control group received lifestyle modifications that are an important part of hypertension management and include weight reduction, following the DASH eating plan with sodium restrictions, daily physical activity, and moderate alcohol consumption. In addition, all patients should be advised to stop smoking to reduce the risk of cardiovascular diseases.
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Other: Relaxation Breathing Exercises Group — This group will preform Relaxation Breathing Exercises that includes Slow Deep Breathing, Pursed lip Breathing, Deep Diaphragmatic Breathing and Alternate Nostril Breathing
  Arms: Relaxation Breathing Exercises Group
Other: Usual Care Group — The control group received lifestyle modifications that are an important part of hypertension management
  Arms: Usual Care Group

SUMMARY:
The objective of this study will be to compare the effects of Relaxation Breathing Exercises on Cardiovascular Parameters among Hypertensive patients. This study will be a Randomized Clinical trial. Data will be collected from Allied and DHQ hospital Faisalabad. One group will receive Breathing Exercises and other group will receive usual care. All subjects will receive a total of three treatment sessions per week over the period of 12 weeks. Outcome will be measured at baseline, 6th and 12th week of treatment.

DETAILED DESCRIPTION:
Hypertension is the leading risk factor for cardiovascular disease and leading cause of premature death globally. Around the world, more than a billion adults suffer with hypertension, which can impact up to 45% of the adult population. All socioeconomic and economic classes experience significant rates of hypertension, and these rates increase with age, reaching up to 60% of people over the age of 60. The Lancet issued a global health survey report in 2010 that included patient data from 67 different countries and identified hypertension as the leading cause of mortality and disability-adjusted life years since 1990. HTN alone accounts for more cardiovascular disease-related deaths in the US than any other modifiable risk factor and is the second-leading preventable cause of death overall, after cigarette smoking. According to recent predictions, there may be up to 1.5 billion hypertensive patients worldwide by 2025, an increase of up to 15%.

Deep breathing exercises involve using a breathing pattern with less than 10 breaths per minute and a lengthy intake period. Benefits of slow, deep breathing exercises include a reduction in pain and stress levels, as well as the management of anxiety and panic. Exercise that involves deep, slow breathing can lower blood pressure, oxygen consumption, metabolism, heartbeat frequency, and frequency of breathing and heartbeat.

Exercises that involve deep breathing can improve vagal tone, stimulate stretch receptors, and lower sympathetic activity. Blood pressure and heart rate are consequently lowered. Shallow breathing increases baroreflex sensitivity and the Vulture-Breuer response, which reduces heart rate and blood pressure.

Diaphragmatic breathing exercises alone have no or little effect. So, the purpose of this study is to combine diaphragmatic breathing exercises with slow deep breathing, alternate nostril breathing and pursed lip breathing to gain its maximum effects and to reduce the stress that is main factor of hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age group: Male and female aged 25 - 45 and above without any other uncontrolled cardiovascular or other diseases, with or without antihypertensive medications.
* Patients who have essential hypertension or stage 1 hypertension.
* SBP between 120 and 139 mmHg
* DBP between 80 - 89 mmHg
* An independent lifestyle should be stable on antihypertensive treatment for a minimum of 2 months before the study and no change in medications during participation in the trial.
* Non-smokers
* None was involved in competitive sports activities

Exclusion Criteria:

* There are signs of secondary hypertension, diabetes mellitus, cardiac disease and pregnancy.
* In use of beta-blockers or centrally acting sympatholytic agents
* 3 or more antihypertensive drugs
* Pregnant women
* Blood pressure greater 180/110 mmHg
* Recent major surgery or admission within 1 year
* Patients with a BMI >30 kg/ m2

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | Baseline; 6th Week; 12th Week
  It is a standard method for measuring exercise capacity in patients with cardiopulmonary disease such as PAH. The 6MWT measures how far a patient can walk in 6 minutes. Walking is an activity performed every day by most patients except for those most severely limited. By assessing patients' ability to exercise, the 6MWT provides a global assessment of respiratory, cardiovascular, neuromuscular, and cognitive function. The 6MWT does not differentiate what limits the patient nor does it assess maximal exercise capacity. Instead, the 6MWT allows the patient to exercise at a daily functional level and is a useful tool for assessing severity of disease, and increasing walk distance correlates with a subjective improvement in dyspnea
Blood Pressure Measurements (SBP & DBP) | Baseline; 6th Week; 12th Week
  An appropriately sized cuff for the arm circumference was installed on the non-dominant arm. Blood pressure was measured every 20 minutes by 24 hours, and awake and sleep periods were determined according to information provided by the patients, the following are 7 strategies recommended by the AHA/AMA for accurate attainment of BP: 1) no conversation, 2) empty bladder, 3) use correct cuff size, 4) place BP cuff on bare arm, 5) support arm at heart level, 6) keep legs uncrossed, and 7) support back and feet

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaltout HA, Eggebeen J, Marsh AP, Brubaker PH, Laurienti PJ, Burdette JH, Basu S, Morgan A, Dos Santos PC, Norris JL, Morgan TM, Miller GD, Rejeski WJ, Hawfield AT, Diz DI, Becton JT, Kim-Shapiro DB, Kitzman DW. Effects of supervised exercise and dietary nitrate in older adults with controlled hypertension and/or heart failure with preserved ejection fraction. Nitric Oxide. 2017 Sep 30;69:78-90. doi: 10.1016/j.niox.2017.05.005. Epub 2017 May 23. PMID 28549665
- [Background] Lebedeva OD, Achilov AA, Mavlyanova ZF, Baranov AV, Achilova SA, Sanina NP, Fesyun AD, Rachin AP, Yakovlev MY, Terentev KV, Reverchuk IV, Velilyaeva AS, Maccarone MC, Masiero S. Is relaxation exercise therapy effective in the management of patients with severe arterial hypertension? Eur J Transl Myol. 2021 Dec 15;31(4):10327. doi: 10.4081/ejtm.2021.10327. PMID 34911289
- [Background] Su TT, Majid HA, Nahar AM, Azizan NA, Hairi FM, Thangiah N, Dahlui M, Bulgiba A, Murray LJ. The effectiveness of a life style modification and peer support home blood pressure monitoring in control of hypertension: protocol for a cluster randomized controlled trial. BMC Public Health. 2014;14 Suppl 3(Suppl 3):S4. doi: 10.1186/1471-2458-14-S3-S4. Epub 2014 Nov 24. PMID 25436830
- [Background] Kundapur R, Modi B, Mary L, Manjula R, Santhosh P, Saxena D. A community-level educational intervention trail to study the impact of life style modification in control of hypertension and diabetes- A non-randomized trial (Before and after intervention study without control). J Family Med Prim Care. 2022 Nov;11(11):6759-6764. doi: 10.4103/jfmpc.jfmpc_2174_21. Epub 2022 Dec 16. PMID 36993009
- [Background] Cherfan M, Vallee A, Kab S, Salameh P, Goldberg M, Zins M, Blacher J. Unhealthy behaviors and risk of uncontrolled hypertension among treated individuals-The CONSTANCES population-based study. Sci Rep. 2020 Feb 5;10(1):1925. doi: 10.1038/s41598-020-58685-1. PMID 32024888